CLINICAL TRIAL: NCT03732846
Title: One-arm, Phase II, Single-center Clinical Study of Anlotinib in the Treatment of Recurrent Small Cell Lung Cancer
Brief Title: Anlotinib in Treatment of Recurrent Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jian Fang, professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTN-SCLC-BCH
Record Dates: First submitted 2018-10-29; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib (Experimental): Take Anlotinib 12mg once daily for two weeks, stop for one week, the program repeats every 21 days until it can not tolerate, or disease progression.
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — Take Anlotinib 12mg once daily for two weeks, stop for one week, the program repeats every 21 days until it can not tolerate, or disease progression

SUMMARY:
Exploring the efficacy and safety of Anlotinib in patients with relapsed small cell lung cancer

DETAILED DESCRIPTION:
This is an one-arm, phase II, single-center clinical study of Anlotinib in the treatment of recurrent small cell lung cancer, the objection is to exploring the efficacy and safety of Anlotinib in patients with relapsed small cell lung cancer.It is going to enroll 43 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Histological or cytologically confirmed small cell lung cancer;
3. Systemic chemotherapy that has previously received at least two or more lines regimen, followed by disease progression or recurrence;
4. According to the RECIST 1.1 standard, there is at least one measurable target lesion;
5. ECOG physical score 0-1 points; expected survival time ≥ 3 months;
6. The main organ function meets the following criteria:

   1. blood routine: absolute value of neutrophils ≥ 1.5 × 109 / L, platelets ≥ 75 × 109 / L, hemoglobin ≥ 80 g / L;
   2. Blood biochemistry: total bilirubin ≤ 1.5 times the upper limit of normal value, aspartate aminotransferase and alanine aminotransferase ≤ 2.5 times the upper limit of normal value (if liver metastasis, ≤ upper limit of normal value 5 times), serum creatinine ≤ 1.5 times the upper limit of normal;
7. Subjects voluntarily joined the study and signed informed consent, with good adherence and follow-up.

Exclusion Criteria:

1. Subjects who have previously used Anlotinib;
2. Systematic anti-tumor treatments have been performed for the past 2 weeks, including chemotherapy, radiotherapy (except for metastatic lesions other than thoracic radiation), targeted therapy, immunotherapy, and biotherapy;
3. Imaging (CT or MRI) shows central tumors in which tumor lesions invade local large blood vessels; imaging (CT or MRI) shows significant pulmonary cavitary or necrotizing tumors; or other factors identified by the investigator that may cause hemoptysis disease;
4. A history of active bleeding within the first 6 months of screening, or receiving thrombolysis or anticoagulant therapy, or the investigator believes that there is a clear tendency to gastrointestinal bleeding (such as esophageal varices with bleeding risk, local activity) Ulcer lesions, etc.) or active hemoptysis;
5. A thrombotic event occurs within 6 months (including arteriovenous thrombosis, pulmonary embolism, cerebrovascular accident, including transient ischemic attack, etc.);
6. Cardiac diseases with obvious clinical symptoms, such as: congestive heart failure, coronary heart disease with obvious symptoms, arrhythmia with difficult drug control (including clinically significant QTc interval prolongation history, or screening period QTc interval women >470ms, Male > 450ms), had myocardial infarction within 6 months, or cardiac insufficiency;
7. Hypertension, which is uncontrolled by the drug, is defined as: systolic blood pressure ≥ 160 mmHg, or diastolic blood pressure ≥ 100 mmHg;
8. Clinically obvious gastrointestinal abnormalities, which may affect the intake, transport or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or patients with total gastrectomy;
9. Surgery (<28 days) before the study was selected or the surgical incision did not completely heal, or there were other unhealed wounds;
10. Active or uncontrolled serious infections;
11. Pregnant or lactating women; those who have fertility are unwilling or unable to take effective contraceptive measures;
12. Increasing the risk associated with participating in a study or study drug, and at the discretion of the investigator, may lead to other conditions in which the patient is not eligible for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-Free survival) | From the date Into this study (signed ICF) to tumor progression or death for any reason, up to 18 months.
  From the date Into this study (signed ICF) to tumor progression or death for any reason.

SECONDARY OUTCOMES:
OS (Overall survival) | From the date Into this study (signed ICF) to death for any reason, up to 18months.
  From the date Into this study (signed ICF) to death for any reason.
DCR (Disease control rate) | From the beginning of treatment, CT and ultrasound examinations are performed every six weeks to assess changes in the disease until the disease progression or death, up to 18 months.
  The rate of CR, PR plus SD
ORR (Objective control rate) | From the beginning of treatment, CT and ultrasound examinations are performed every six weeks to assess changes in the disease until the disease progression or death, up to 18 months.
  The rate of CR and PR

CONTACTS AND LOCATIONS:
Overall Officials: Jian Fang, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided